CLINICAL TRIAL: NCT05208671
Title: Nutrition to Optimize, Understand, and Restore Insulin Sensitivity in HIV for Oklahoma
Acronym: NOURISH-OK
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oklahoma (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 12509; 5R01DK127464 (NIH)
Record Dates: First submitted 2022-01-11; First posted 2022-01-26 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2024-04

CONDITIONS: HIV; Insulin Resistance; Food Insecurity
Keywords: food as medicine; nutrition
MeSH Terms: conditions — Insulin Resistance

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NOURISH Food Box (Experimental): 12-week food assistance with low Dietary Inflammatory Index (DII) foods
  Interventions: Other: NOURISH Food Box
- Wait-list Control (No Intervention): Wait-list control group eligible to receive NOURISH box after study period

INTERVENTIONS:
Other: NOURISH Food Box — Selection of healthy groceries designed to reduce chronic inflammation and improve insulin resistance with healthy cooking/self-care curriculum
  Arms: NOURISH Food Box

SUMMARY:
The NOURISH-OK Study will identify how food insecurity contributes to insulin resistance, an important surrogate marker of many co-morbidities in HIV disease, using an integrated framework to identify key leverage points for insulin resistance. Drawing from these pathways, this study will adapt and evaluate a community-driven, science-informed "food as medicine" intervention designed to lower insulin resistance through healthy food access, food utilization skills, and other self-care behaviors. Knowledge gained from this study can benefit those living with HIV through the prevention and more effective management of pre-diabetes, diabetes, obesity, and non-alcoholic fatty liver disease.

DETAILED DESCRIPTION:
The community-based participatory research study will be conducted in Oklahoma, and include HIV-positive individuals living in urban and rural communities. The first two aims are observational, the third aim will test an intervention.

Aim 1: Test and refine a conceptual integrated framework of food insecurity and insulin resistance to identify significant structural, social, behavioral, and biological pathways as candidate intervention points. This aim will be accomplished using a cross-sectional survey (n=410 final sample size) and a one-month observational sub-study from the main study sample (n=89 final sample size) to collect intensive measures of dietary intake and gut microbiome samples.

Aim 2: Adapt a home-delivered grocery and cooking self-care NOURISH-OK intervention to address key nutrition disparities and other health risk behaviors identified as significant path contributors to insulin resistance among people living with HIV. This aim will be achieved through a series of interviews and focus groups with people living with HIV who are food insecure (n=45 qualitative study subjects, including interviews and focus groups).

Aim 3: Implement the 12-week NOURISH-OK intervention and assess it for feasibility, acceptability, and preliminary impact using a randomized wait-list control design (n=234). This study will use a simple randomized wait-list control trial design. Additionally, the investigators will invite a random selection from the main study sample (n=80) to participate in more intensive data collection, including multiple 24-hr food recalls and stool samples during the intervention period to assess for food insecurity, dietary, and gut microbiome changes throughout the intervention periods.

ELIGIBILITY:
Inclusion Criteria:

* HIV-positive with income <400% federal poverty level
* at least 1 risk factor for insulin resistance per the National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (i.e., overweight/obesity, age 45 yrs or older, immediate family member with diabetes, non-white race, physical inactivity, history of gestational diabetes, history of heart disease or stroke, diagnosis of polycystic ovarian syndrome, high blood pressure, high cholesterol, or hepatitis C virus antibody positivity
* using antiretroviral therapy for at least 6 months
* English-speaking

Exclusion Criteria:

* participating in another health-related research study
* receiving treatment for a terminal or other serious illness, such as cancer or end-stage renal failure
* plan to move outside of Oklahoma during the study period
* does not have an address that can accept home-delivered groceries

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 234 (Estimated)
Dates: Start 2020-10-09 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Change from baseline insulin sensitivity at 12-weeks | Baseline; 12-weeks
  Quantitative Insulin-Sensitivity Check Index (QUICKI)

SECONDARY OUTCOMES:
Change from baseline food security at 6-weeks, 12-weeks, and 16-weeks | Baseline; 6-weeks; 12-weeks; 16-weeks
  10-item US Adult Food Security Module (0-10 point range; higher score reflects lower food security)
Change from baseline dietary intake at 6-weeks, 12-weeks, and 16-weeks | Baseline; 6-weeks; 12-weeks; 16-weeks
  Dietary Inflammatory Index (DII) (higher score reflects diet with greater inflammatory potential)
Change from baseline skin carotenoid at 12-weeks | Baseline; 12-weeks
  reflection spectroscopy using "Veggie Meter" device (higher score reflects higher carotenoid status)
Change from baseline chronic inflammation at 12-weeks | Baseline; 12-weeks
  C-reactive protein (blood measure) (higher score reflects higher chronic inflammation)

OTHER OUTCOMES:
Change from baseline gut microbiome composition at 12-weeks | Baseline; 12-weeks
  Microbiome composition (diversity) - subsample only

CONTACTS AND LOCATIONS:
Overall Officials: Marianna S Wetherill, PhD, MPH, RD, Principal Investigator — University of Oklahoma
Locations (1):
- OU Integrative Immunology Center, Tulsa, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, ICF
Time Frame: Made available within 12 months of study end.
Access Criteria: Written request to PI.

REFERENCES:
- [Derived] Wetherill MS, Bakhsh C, Caywood L, Williams MB, Hartwell ML, Wheeler DL, Hubach RD, Teague TK, Kohler G, Hebert JR, Weiser SD. Unpacking determinants and consequences of food insecurity for insulin resistance among people living with HIV: Conceptual framework and protocol for the NOURISH-OK study. Front Clin Diabetes Healthc. 2022;3:947552. doi: 10.3389/fcdhc.2022.947552. Epub 2022 Aug 16. PMID 36225538
- See also: NOURISH-OK Study Information Webpage — http://www.tulsacares.org/nourish/